CLINICAL TRIAL: NCT00389246
Title: Evaluation of Consultation Including Genetic Aspects of Obesity
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Winfried Rief, Professor Dr., Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WR001; 01GP0209
Record Dates: First submitted 2006-10-17; First posted 2006-10-18 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Obesity
Keywords: obesity; genetic consultation; randomized controlled trial
MeSH Terms: conditions — Obesity | interventions — Referral and Consultation

INTERVENTIONS:
Behavioral: Consultation without genetic information
Behavioral: Consultation with genetic information

SUMMARY:
More than 1,000 obese people are screened for genetic mutations (MC4R). Those with positive screenings as well as 320 randomly selected people without MC4R mutations are randomized to 2 consultation types: one including recommendations for eating and physical activity behavior, the other with an additional part on genetic determinants and actions in obesity. It is hypothesized that obese people with obesity-specific genetic mutations, and obese people with a family history of obesity, benefit more if the consultation includes additional elements on genetic determinants.

DETAILED DESCRIPTION:
More than 1,000 obese people are screened for genetic mutations (MC4R). Those with positive screenings as well as 320 randomly selected people without MC4R mutations are randomized to 2 consultation types: one including recommendations for eating and physical activity behavior, the other with an additional part on genetic determinants and actions in obesity. Their results are compared to a control group (n>100). It is hypothesized that obese people with obesity-specific genetic mutations, and obese people with a family history of obesity, benefit more if the consultation includes additional elements on genetic determinants.

The following variables are used: BMI, SCID interview for mental disorders, Stunkard's body silhouttes for participants and their parents and siblings, Restraint Eating Scale, PANAS, Well-being scale, body acceptance, shame and guilt, coping with obesity, participant's satisfaction with consultation.

Assessment Points: before consultation, after consultation, 6 months later.

ELIGIBILITY:
Inclusion Criteria:

* BMI > 30

Exclusion Criteria:

* Brain damage

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420
Dates: Start 2002-09; Study Completion 2005-06

PRIMARY OUTCOMES:
Feeling guilty for being overweight
Negative affectivity
Self-control

SECONDARY OUTCOMES:
weight
body acceptance
restraint eating
qualityof life
coping

CONTACTS AND LOCATIONS:
Overall Officials: Winfried Rief, PhD, Principal Investigator — Philipps University of Marburg, Marburg, Germany

REFERENCES:
- See also: Philipps University of Marburg, Germany — http://www.uni-marburg.de